CLINICAL TRIAL: NCT00470938
Title: A Randomized Controlled Trial of the Effects of Reactive Neuromuscular Training on Balance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Kristan Giggey, DC, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RD0202070062
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Balance

INTERVENTIONS:
Device: SpineForce Reactive Neuromuscular Trainer

SUMMARY:
Falls are a major concern for the geriatric population and represent a significant public health problem. Various interventions are being explored to improve balance and decrease falls in the elderly. Success has been shown in some programs; various exercise interventions place emphasis on strength, balance, or endurance exercises. Results reported in the literature are still equivocal. Controversy exists as to optimal types of exercise, and the optimum frequency, duration, and intensity of exercise. It is believed that the SpineForce device, which places a unique combination of strength and balance demands upon the user, can result in rapid increases in balance as compared to other rehabilitation programs. Gains in balance have implications for geriatric populations as well as those seeking enhanced sports performance and injury prevention. The Purpose of this study is to assess the SpineForce device as a novel intervention in the treatment of balance disorders.

ELIGIBILITY:
Inclusion Criteria:

* Young, healthy adults between the ages of 20 - 30, asymptomatic with respect to any balance specific disorder, and who are currently enrolled at Logan College.

Exclusion Criteria:Exclusion criteria include:

* A previous lower extremity injury;
* Previous lower extremity surgery;
* A visual or vestibular condition with accompanying balance difficulty;
* A diagnosis of Knee osteoarthritis;
* Currently receiving spinal manipulative therapy;
* Current participation in a regular exercise program;
* Use of any prescription medication, or herbal substance that may affect balance;
* Pregnancy

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodger Tepe, PhD, Study Director — Logan College of Chiropractic